CLINICAL TRIAL: NCT05320146
Title: A Phase 1b, Open-Label Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Adult Patients With Presumed Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Sub Study of the Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Patients With Presumed Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Type: Observational
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CORT118335-861 - Sub Study
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Nonalcoholic Steatohepatitis; NASH; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and Serum samples will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CORT118335-860 Participants: This group will include patients who participated in CORT118335-860 study and received at least one dose of miricorilant.
  Interventions: Other: MRI-PDFF
- CORT118335-861 Participants: This group will include patients who participated in CORT118335-861 study and received at least one dose of miricorilant.
  Interventions: Other: MRI-PDFF

INTERVENTIONS:
Other: MRI-PDFF — Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) is a MRI-based diagnostic imaging biomarker of the liver.

SUMMARY:
This optional sub study is a part of the phase 1b, Open-Label Study is to assess the safety, efficacy of miricorilant in patients with presumed Nonalcoholic Steatohepatitis (NASH)

DETAILED DESCRIPTION:
This optional sub study is a part of the phase 1b, Open-Label Study is to assess the safety, efficacy of miricorilant in patients with presumed Nonalcoholic Steatohepatitis (NASH).

All patients who participated in the current study (CORT118335-861) or the Corcept Phase 2a NASH study (CORT118335-860), and who received at least one dose of miricorilant will be eligible for participation in an observational follow-up study; this includes patients who either terminated early or are study completers.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in either Study CORT118335-861 (current study) or Study CORT118335-860 (Corcept Phase 2a NASH study) and received at least one dose of miricorilant; this includes patients who terminated early from the study or completed the study.
* Have not participated in any other clinical trial following study completion in either Study CORT118335-861 or Study CORT118335-860.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that have previously enrolled in CORT118335-860 or in CORT118335-861 and have received at least one dose of miricorilant.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change in liver-fat content assessed by MRI-PDFF after the last dose of study drug. | Baseline Day 1 up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (9):
- United States (9):
  - Site 207, Chandler, Arizona
  - Site 209, Tucson, Arizona
  - Site 214, Panorama City, California
  - Site 233, Santa Ana, California
  - Site 211, Austin, Texas
  - Site 213, Edinburg, Texas
  - 305, Houston, Texas
  - Site 212, San Antonio, Texas
  - 226, Seattle, Washington

REFERENCES:
- See also: Clinical Trial public posting for CORT113885-860 — https://clinicaltrials.gov/ct2/show/NCT03823703
- See also: Clinical Trial public posting for CORT118335-861 — https://clinicaltrials.gov/ct2/show/NCT05117489